CLINICAL TRIAL: NCT02359240
Title: Skeletal Muscle Wasting in Patients With Sepsis
Brief Title: HO-1 and Muscle Mitochondrial Dysfunction in Sepsis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Xiaoming Deng, Chief, Professer, Changhai Hospital
Other Study IDs: CH1502
Record Dates: First submitted 2015-01-28; First posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Sepsis; Atrophy
MeSH Terms: conditions — Sepsis; Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — skeletal muscle
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- sepsis: Patients with a diagnosis of sepsis or severe sepsis,immobilization for 3 days at least. Therapy according to the SSC guidelines will be applied. therapy according to SSC guidelines and muscle biopsy
  Interventions: Procedure: therapy according to SSC guidelines and muscle biopsy
- Patients with femoral fractures: non septic patients with a femoral fracture,who need an fixation surgery.standard surgery for femoral fracture and muscle biopsy will be performed.
  Interventions: Procedure: standard surgery for femoral fracture and muscle biopsy

INTERVENTIONS:
Procedure: therapy according to SSC guidelines and muscle biopsy — Septic patients will be treated according to the international guidelines for management of severe sepsis and septic shock 2012. Skeletal muscle biopsies, blotted free from blood, are frozen within 30 seconds in liquid nitrogen, and stored in liquid nitrogen until processing.150-300 mg muscle (wet weight) was routinely obtained , which is more than sufficient for the analyses proposed, with some muscle remaining for any additional validation assays that may arise during the course of the research. Muscle will be processed either for isolation of mRNA/microRNA or protein
  Groups: sepsis
Procedure: standard surgery for femoral fracture and muscle biopsy — Patients with femoral fracture will under standard surgery for fracture fixation. Percutaneous needle muscle biopsies will be performed. Skeletal muscle biopsies, blotted free from blood, are frozen within 30 seconds in liquid nitrogen, and stored in liquid nitrogen until processing.150-300 mg muscle (wet weight) was routinely obtained , which is more than sufficient for the analyses proposed, with some muscle remaining for any additional validation assays that may arise during the course of the research. Muscle will be processed either for isolation of mRNA/microRNA or protein
  Groups: Patients with femoral fractures

SUMMARY:
The current project was designed to examine dynamic changes in muscle wasting during sepsis. Researchers will focus the mitochondrial dysfunction of muscle cells and investigate the role of HO-1 in it. Researchers interested in identifying factors involved in the pathology of muscle wasting during sepsis.

DETAILED DESCRIPTION:
Rapid muscle atrophy or muscle wasting occured to septic patients.Sepsis induced muscle wasting has become a severe, frequent, and persistent complication among critically ill patients. Multiple factors including ubiquitin-proteasome system, proinflammatory cytokines and oxidative stress contribute muscle proteolysis.

It is known that heme oxygenase-1 (HO-1) possesses a variety of functions like anti-inflammatory, antioxidative and anti-apoptosis effects. In order to investigate the mechanisms under the condition, researchers are going to examine the role of HO-1 in muscle atrophy during sepsis.

ELIGIBILITY:
Inclusion Criteria:

* sepsis, severe sepsis, septic shock
* clinical reason for fixation surgery of femoral fractures

Exclusion Criteria:

* no informed consent
* medical history of myopathy
* unintended weight loss before surgery or ICU admission
* chronic use of corticosteroids

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: septic patients; non septic patients with a femoral fracture,who need an fixation surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
HO-1 mRNA and protein expression, mitochondria function of musculus vastus lateralis | 3 days after diagnosis

SECONDARY OUTCOMES:
length of ICU stay | 60 days
length of mechanical ventilation | 60 days
muscle myosin content | 3 days after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Deng, M.D., Ph.D., Principal Investigator — Changhai Hospital
Locations (1):
- Anesthesiology and Intensive Care, Changhai Hospital, Shanghai, Shanghai Municipality, China